CLINICAL TRIAL: NCT05366790
Title: Application of a Brief Digital Screening Tool to Address Parental and Adolescent Tobacco and Electronic Cigarette Use in Pediatric Medical Care (CanCEASE) - a Pilot Study
Brief Title: A Brief Digital Screening Tool to Address Tobacco and E-cigarette Use in Pediatric Medical Care
Acronym: CanCEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Olivier Drouin, M.D., M.Sc M.P.H., Pediatrician and Clinical Assistant Professor, Departments of Paediatrics and Department of Social and Preventive Medicine, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 470909
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Tobacco Use; Tobacco Cessation; Second Hand Tobacco Smoke; Smoking, Tobacco; Vaping
Keywords: Smoking cessation; second hand smoke; nicotine replacement therapy; vaping; adolescents
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation; Tobacco Smoking; Vaping; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to received either the CEASE intervention (supportive smoking cessation services) or care as usual.
Who Masked: Investigator
Masking Description: Investigators will be blinded to the participants' group allocation. In this pragmatic trial, pediatricians may decide to discuss smoking and/or vaping with families as part of their usual care, and participants may mention the CEASE/CEASE-A intervention during the encounter with the provider. As such, participants and physicians will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEASE Intervention arm (Experimental): The CEASE and CEASE-A interventions are tobacco and vaping cessation interventions delivered in pediatric practices, leveraging existing healthcare and community resources. They integrate evidence-based tobacco use screening and cessation assistance into routine visits to pediatric clinics. CEASE and CEASE-A are based on the 5A's model of smoking cessation: Ask about smoking, Advise to quit, Assess readiness to quit, Assist with a quit plan and Arrange follow-up. Given that CEASE and CEASE-A are one-time interventions, "Arrange" is removed, and the fourth step "Assist" is divided into two parts: a) providing phone/text/app quit support and b) providing NRT.
  CEASE-A follows the same format at CEASE, but is modified slightly to address smoking and vaping in the adolescent target population
  Interventions: Behavioral: CEASE and CEASE-A
- Control: Usual care condition (No Intervention): The control condition will be care as is usually delivered in participating clinics with the possibility of receiving direct linkage with cessation services delivered via CEASE/CEASE-A at the end of the 6-month study period. Current practice does not include routine provision of assistance for parental/adolescent smoking or e-cigarette cessation (e.g., referral to quitlines, NRT prescription).

INTERVENTIONS:
Behavioral: CEASE and CEASE-A — CEASE (for parents) and CEASE-A (for adolescents) are evidence-based tobacco and vaping cessation interventions delivered in pediatric practices.
  Arms: CEASE Intervention arm

SUMMARY:
Tobacco use is the single greatest preventable cause of morbidity and mortality in Canada, accounting for 48,000 deaths and $16.2 billion annually in attributable health-related costs. Parents who smoke are often medically underserved and visit their child's doctor more than their own; 25% of all adult smokers have children seen in child healthcare. When parents quit smoking, their life expectancy is increased by more than 10 years, tobacco-related poor pregnancy outcomes are eliminated, children's risk of becoming smokers decreases 4-fold, families have more money for necessities, and children are less likely to suffer from diseases caused by tobacco smoke exposure.

Despite free tobacco cessation services in every province and widespread insurance coverage of NRT, parental tobacco screening and cessation support rarely happens in pediatric care, thus there is potential for major health benefits from a routinely delivered tobacco control program to parents in this setting.

The investigators will conduct a 12-month single centre, pragmatic, single-blind pilot RCT of CEASE vs. usual care of 70 parents who use cigarettes and/or vaping products whose children are seen in pediatric clinics at the CHU Sainte-Justine. A similar trial, CEASE-A will be conducted with 70 adolescents ages 14-17.

Objectives:

1. Perform a pilot RCT of the Clinical Effort Against Secondhand Smoke (CEASE) intervention in Canada. CEASE is an evidence-based parental smoking cessation intervention to ensure that every parent who uses cigarettes and/or nicotine vaping products and visits their child's pediatrician receives nicotine dependence treatment
2. Conduct an ancillary pilot RCT of CEASE-A to deliver evidence-based support for adolescents who use tobacco and/or nicotine vaping products Outcomes include pilot process outcomes and preliminary effectiveness outcomes to assess feasibility and inform the preparation of a future large-scale RCT.

This pilot RCT will provide the data necessary to plan a fully powered RCT assessing the effectiveness of CEASE and CEASE-A for smoking and vaping cessation.

DETAILED DESCRIPTION:
Background: Tobacco use is the single greatest preventable cause of morbidity and mortality in Canada, accounting for 48,000 deaths and $16.2 billion in attributable health-related costs annually. Twenty-five percent of all adult smokers have children who are seen in child healthcare offices. When parents quit smoking, their life expectancy is increased by more than 10 years, tobacco-related poor pregnancy outcomes are eliminated, children have 4-fold lower risk of becoming smokers, families have more money for necessities, and children are less likely to suffer from diseases caused by tobacco smoke exposure. Parents who smoke are often medically underserved and visit their child's doctor more than their own. Thus, a routinely delivered tobacco control program to parents in the pediatric context would provide a major health benefit to the nation. Yet, parental tobacco screening and cessation support happens less than 5% of the time in pediatric practices despite free tobacco cessation quitlines and services in every province and widespread insurance coverage of nicotine replacement therapy (NRT).

Specific Objectives:

Primary objective:

• Perform a pilot randomized controlled trial (RCT) of the Clinical Effort Against Secondhand Smoke (CEASE) intervention in Canada. CEASE is an evidence-based parental smoking cessation intervention to ensure that every parent who uses cigarettes and/or nicotine vaping products and visits their child's pediatrician receives nicotine dependence treatment.

Secondary objective:

• Conduct an ancillary pilot RCT of CEASE-A, an extension of CEASE, to deliver evidence-based support for adolescents who use tobacco and/or nicotine vaping products.

These pilot RCTs will inform whether full scale RCTs of CEASE/CEASE-A are feasible.

Design: The investigators will conduct a 12-month single centre, pragmatic, single-blind pilot RCT of the CEASE intervention vs. care as usual (ratio 1:1) of 70 parents who use cigarettes and/or vaping products whose children are seen in pediatric clinics at the CHU Sainte-Justine. A similar trial will be conducted with 70 adolescents ages 14-17 with the CEASE-A intervention.

Population: For the primary objective, the population will be parents of children 0-17 years old and who use tobacco or nicotine vaping products. "Users" will be defined as those answering "Yes" to the screening question: "Have you smoked a single cigarette or used nicotine vaping products, even a puff, in the past 7 days?"

For the secondary objective (CEASE-A), the population will be adolescent patients aged 14-17 years who use tobacco or nicotine vaping products. "Adolescent users" will be defined as those answering "Yes" to the screening question: "Have you smoked a single cigarette or used a nicotine vaping product, even a puff, in the past 7 days?"

Intervention: The CEASE intervention is a parental tobacco and vaping cessation intervention delivered in pediatric practices, leveraging existing healthcare and community resources. It integrates evidence-based tobacco use screening and cessation assistance into routine visits to pediatric clinics. CEASE is based on the 5A's model of smoking cessation: Ask about smoking, Advise to quit, Assess readiness to quit, Assist with a quit plan and Arrange follow-up. Given that CEASE is a one-time intervention, "Arrange" is removed, and the fourth step "Assist" is divided into two parts: a) providing phone/text/app quit support and b) providing NRT.

CEASE-A follows the same format at CEASE, but is modified slightly to address smoking and vaping in the adolescent target population

Control: The control condition will be care as is usually delivered in participating clinics with the possibility of receiving direct linkage with cessation services delivered via CEASE/CEASE-A at the end of the 6-month study period. Current practice does not include routine provision of assistance for parental/adolescent smoking or e-cigarette cessation (e.g., referral to quitlines, NRT prescription).

Follow-up includes three data collection time points at 1-, 3- and 6-months after recruitment.

Outcomes

Outcomes will include pilot process (feasibility) outcomes to ensure a large RCT is feasible, as well as preliminary effectiveness outcomes to inform the preparation of a future large-scale RCT.

Pilot RCT process outcomes:

1. Parental and adolescent recruitment rates

   * Number of potential participants (parent, adolescent) per month for each clinic
   * Proportion of potential participants screened for eligibility
   * Self-reported smoking and vaping rates among parents and adolescents screened
   * Number of eligible parents and adolescents per month for each clinic
   * Proportion of eligible participants approached who are enrolled in the study
   * Reasons for declining participation in the study
   * Number of participants recruited per month (parents and adolescents)
2. Feasibility of the intervention

   * Proportion of eligible participants in each category (parents and adolescents) who declare interest in smoking/vaping cessation
   * Proportion of eligible participants (parents and adolescents) who want to be connected with smoking/vaping cessation services (quitlines)
   * Proportion of eligible participants in each category who want to receive NRT
3. Protocol fidelity

   * Proportion of participants who complete the baseline questionnaire
   * Proportion of participants who want to be connected to quitlines who are referred i. Proportion of participants who received a communication from the quitlines at 1 month
   * Proportion of participants who want to receive NRT who receive a prescription i. Proportion of participants who have used NRT 1 month later
4. Study retention and completion of follow-up questionnaires

   * Proportion of participant that drop out or are lost to follow-up at 1, 3 and 6 months
   * Availability of self-reported smoking/vaping status at 1-, 3- and 6-month
   * Complete data available (1-, 3- and 6-month surveys) for retained participants
   * Availability of cotinine-testing at 1-, 3- and 6 months
5. Minimal interruption of clinic workflow

   * Average weekly and monthly patient volumes in each clinic
   * Key informant interviews or written survey with front desk staff, and clinical staff to document impacts of the intervention on clinic workflow.

Effectiveness outcomes

* Abstinence at 6 months: % of parental/adolescent users who report 7-day abstinence at 6-month follow-up. We will collect self-reported smoking and vaping status using the validated single items "Have you smoked a single cigarette, even a puff, in the past 7 days?" and "Have you used a nicotine vaping product, even a puff, in the past 7 days?"
* Cotinine-confirmed quit: Participants who self-report 7-day abstinence at 1, 3 and/or 6 months will receive a sampling kit by mail along with instructions on how to collect the urine for biochemical confirmation of smoking/vaping cessation

Secondary effectiveness outcomes

* Intent to quit smoking and/or vaping at recruitment and follow-up
* Quit attempts at 1-, 3- and 6- months

Statistical plan and sample size calculation:

For this pilot RCT, process outcomes will be examined using descriptive statistics and compared between intervention and control groups using chi-square tests.

Sample size calculation To estimate participation rate, using a sample size of 70 participants per age group will allow for a 95% confidence interval within 15% of the estimate obtained. As such, if participation rate in the feasibility study of 60% is observed, the 95% C.I. would be (44.2%, 75.8%). As recruitment rates may differ between adult and adolescent participants, the investigators will enroll 70 parents and 70 adolescents for this pilot study to obtain two participation rates estimates.

Relevance The proposed pilot RCT will provide the data necessary to plan a fully powered RCT assessing the effectiveness of CEASE and CEASE-A for smoking and vaping cessation. It will also help test this evidence-based intervention in a new population, adolescents, with high potential to act early in the life course and meaningfully reduce the societal burden associated with tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legal guardians of children 0-17 years old and who smoke or use nicotine vaping products. "User" will be defined as those who answer "Yes" to the screening questions:

  * "Have you smoked a single cigarette, even a puff, in the past 7 days?" (smoking);
  * "Have you used an e-cigarette or vaping device containing nicotine, even a puff, in the past 7 days? (vaping).

For CEASE-A, adolescent patients aged 14-17 years who smoke or use nicotine vaping products will be considered. "Adolescent User" will be defined by those who answer "Yes" to the same screening question as parents.

Parents will be eligible if 1) they are at least 18 years old, 2) their child is 0-17 years of age, 3) are attending a regular scheduled medical appointment, and 4) are sufficiently proficient in either French or English (able to read and answer a written questionnaire).

Adolescents will be eligible if they are 14-17 years-old, meet criteria 3) and 4) above, and have provided informed consent (in Québec, adolescents aged 14 years can provide consent). Adolescents whose parent(s) (if present) are not agreeable to their participation will be excluded.

Exclusion Criteria:

* Families presenting to the clinic without a scheduled medical appointment will be excluded. There will be no other exclusion criteria.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Parental and adolescent recruitment rates | 12 months of study follow up
  The proportion of eligible participants approached who are enrolled in the study. Number of participants recruited per month.
Feasibility of the intervention | 12 months of study follow up.
  Proportion of eligible participants in each category (parents and adolescents) who declare interest in smoking/vaping cessation, who wish to be connected with smoking/vaping cessation services (quitlines), and who want to receive NRT.
Protocol fidelity | 6 months of participant follow up.
  Proportion of participants who complete the baseline questionnaire, proportion of participants who want to be connected to quitlines who are referred, and proportion who want to receive NRT and receive a prescription.
Study retention and completion of follow-up questionnaires | 6 months of participant follow up.
  Proportion of participant that drop out or are lost to follow-up at 1, 3 and 6 months
  * Availability of self-reported smoking/vaping status at 1-, 3- and 6-month
  * Complete data available (1-, 3- and 6-month surveys) for retained participants
  * Availability of cotinine-testing at 1-, 3- and 6 months
Abstinence at 6 months | 6 months of participant follow up.
  % of parental/adolescent users who report 7-day abstinence at 6-month follow-up. We will collect self-reported smoking and vaping status using the validated single items "Have you smoked a single cigarette, even a puff, in the past 7 days?" and "Have you used a nicotine vaping product, even a puff, in the past 7 days?"
Cotinine-confirmed quit | 6 months of participant follow up.
  Participants who self-report 7-day abstinence at 1, 3 and/or 6 months will receive a sampling kit by mail along with instructions on how to collect the urine for biochemical confirmation of smoking/vaping cessation

SECONDARY OUTCOMES:
Proportion of participants reporting intent to quit smoking/vaping | 6 months of participant follow-up
  Participant self-reported intention to quit smoking and/or vaping at recruitment and follow-up
Proportion of participant reporting quit attempts at 1-, 3- and 6- months | 6 months of participant follow-up
  Participant self-reported smoking or vaping cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Drouin, MD, MSc MPH, Principal Investigator — CHU Sainte-Justine Research Centre; Nicholas Chadi, MD, MPH, Principal Investigator — CHU Sainte-Justine Research Centre
Locations (1):
- Pediatric Clinic of the CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chadi N, Diamant E, Perez T, Al-Saleh A, Sylvestre MP, O'Loughlin J, Winickoff JP, Drouin O. A Brief Digital Screening and Intervention Tool for Parental and Adolescent Tobacco and Electronic Cigarette Use in Pediatric Medical Care in Canada: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 30;12:e47978. doi: 10.2196/47978. PMID 38032712